CLINICAL TRIAL: NCT06897358
Title: A Study to Assess Safety and Tolerability, and Explore Efficacy of Leniolisib for Immune Dysregulation in Common Variable Immunodeficiency (CVID)
Brief Title: Leniolisib for Immune Dysregulation in CVID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Collaborators: Lahey Hospital & Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE 8201
Record Dates: First submitted 2025-03-12; First posted 2025-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Common Variable Immunodeficiency (CVID)
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — leniolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leniolisib (Experimental): All subjects participating will receive leniolisib film-coated tablets (FCTs) with a planned dose regimen consisting of a starting dose of 10 mg twice daily (BID) for 4 weeks, followed by a dose escalation to 30 mg BID for 4 weeks, and then 70 mg BID for an additional 16 weeks.
  Interventions: Drug: Leniolisib

INTERVENTIONS:
Drug: Leniolisib — Planned dose will range from 10 mg twice daily to 70 mg twice daily
  Other Names: Joenja

SUMMARY:
In this study, common variable immunodeficiency (CVID) patients will all receive the study drug, leniolisib, for a treatment period of 6 months. Participants will start on a lower dose of leniolisib, followed by a mid and then a higher dose level. The primary goal is to assess the safety and tolerability of leniolisib, and secondary goal is to assess the potential for leniolisib to provide benefits for patients.

DETAILED DESCRIPTION:
The study includes administration of increasing dose levels of leniolisib in approximately 20 CVID patients presenting with clinical manifestations of immune dysregulation at study entry. Enrollment will include both patients without and those with genetic drivers identified for their CVID.

All subjects participating will receive leniolisib film-coated tablets (FCTs) with a planned dose regimen consisting of a starting dose of 10 mg twice daily (BID) for 4 weeks, followed by a dose escalation to 30 mg BID for 4 weeks, and then 70 mg BID for an additional 16 weeks. Dose adjustments are allowed during treatment if deemed clinically necessary.

Subjects not continuing leniolisib treatment outside the current protocol will be followed up, with the EoS visit planned to occur approximately 28 days after last dose of leniolisib.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 12 to 75 years of age (inclusive).

   a. Specifically at sites located in the United Kingdom subjects must be 18 to 75 years of age (inclusive)
2. Subject must have a minimum body weight of 45 kg
3. Subject has a clinical diagnosis of CVID supported by all of the following (a thru c):

   1. A low IgG level compared to age-adjusted reference range [OR if this cannot be documented, subject must have one of the following: i) absent isohemagglutinins and/or poor response to vaccines; or ii) Low class-switched memory B cells less than 2%]
   2. Low IgA and/or IgM compared to age-adjusted reference range
   3. No identified secondary causes of hypogammaglobulinemia
4. Inborn Errors of Immunity/ PID Panel testing:

   1. Lacks an identified pathogenic/likely pathogenic genetic driver for their CVID primary immunodeficiency OR
   2. Subject has an identified pathogenic/likely pathogenic genetic driver(s) for their CVID limited to the following genes: TNFRSF13B (TACI), TNFRSF13C (BAFFR), CD19, CD20, CD81, CR2 (CD21), LRBA, CTLA4, NFKB1, NFKB2, IKZF1 (excluding variants associated with combined immune deficiency), CARD11 (gain of function), SH3KBP1, SEC61A1 IRF2BP2, CTNNBL1, TWEAK or PTEN.
5. Subject has lymphoproliferation, as evidenced by CT imaging: splenomegaly with craniocaudal spleen measurement >10 cm and/or lymphadenopathy with at least 1 measurable index lymph node (long axis >1.5 cm) as per Cheson methodology.
6. Subject has at least ONE of the following CVID clinical manifestations of immune dysregulation:

   1. Clinical symptoms related to splenomegaly or lymphadenopathy which interfere with activities of daily living or are associated with chronic pain, dyspnea, functional impairment, or limitations in usual activities
   2. One or more blood cytopenias related to CVID (and not due to other medical conditions such as iron-deficiency or lead exposure) defined as hemoglobin <10 g/dL, platelet count <100,000/µL, and/or neutrophil count <1,000/µL
   3. Previous pathologic confirmation of ILD and attributed to CVID by the Investigator with quantifiable CT chest imaging findings evident on baseline CT scan
   4. Clinical diagnosis of CVID enteropathy or other GI tract diagnosis attributable to CVID by the Investigator which involves the small intestine and meets the following enteropathy criteria:

   i. Clinical symptoms of GI disease including at least 1 of: abdominal pain or diarrhea at least 3 days of the week for at least 4 weeks or longer, or dependence on supplemental enteral or parenteral nutrition ii. Lacks a clinical diagnosis of Celiac Disease, and negative human leukocyte antigen (HLA)-DQ2 and -DQ8 testing at screening iii. Presence of small bowel villous shortening/atrophy/blunting with or without intraepithelial lymphocytosis noted in a pathology report pertaining to a small bowel biopsy performed within 5 years of enrollment iv. Negative stool PCR Gastrointestinal Profile at screening
7. At screening, vital signs. Ranges:

   Systolic blood pressure 80-159 mm Hg Diastolic blood pressure 50-109 mm Hg Pulse rate 50-110 beats per minute (bpm) Oxygen saturation 93-100%
8. Subjects or their legal representatives (for subjects under the age of 18 years) must be able to communicate with the Investigator and understand and comply with the requirements of the study, including an ability to provide written informed consent.

Exclusion Criteria:

1. Laboratory evidence of significant T cell deficiency including CD4+ T cells <200/uL.
2. Laboratory evidence of significant NK cell deficiency including NK cells <1% of peripheral blood lymphocytes or less than 50/mcL.
3. Clinical history of infections suggestive of clinically significant T cell or NK cell deficiency such as Pneumocystis jirovecii, atypical mycobacteria, severe warts, or unusually severe (as determined by the PI) infections with herpesviruses.
4. Presence of uncontrolled chronic/recurrent infectious disease (except those considered to be characteristic of antibody deficiency).
5. Positive blood polymerase chain reaction (PCR) for cytomegalovirus.
6. Evidence of tuberculosis infection
7. Positive blood cryptococcal antigen
8. Previous or concurrent use of immunosuppressive medication, such as:

   * Use of an mTOR inhibitor or a PI3K inhibitor within 3 weeks.
   * Rituximab or other B cell depleting antibodies, belimumab, cyclophosphamide, or alemtuzumab within 6 months.
   * Cyclosporine A, mycophenolate mofetil, 6-mercaptopurine, azathioprine, methotrexate, tacrolimus, ruxolitinib, or other Janus kinase (JAK) inhibitors within 3 weeks.
   * Glucocorticoids above 25 mg prednisone or equivalent per day within 2 weeks
   * Immunosuppressive monoclonal or polyclonal antibody therapeutics such as directed against TNF-alpha, α₄β₇ integrin, IL-6, IL-12/IL-23 and others within 5 half-lives
   * Other immunosuppressive agents expected to have a significant impact on immune cell number or function.
   * Abatacept is allowed during study if the subject has been receiving a stable dosing regimen for more than 3 months .
   * Enteral budesonide is allowed during study if the subject has been receiving a stable dosing regimen for more than 3 months.
9. Subject is receiving concurrent treatment with another investigational therapy or use of another investigational therapy less than 4 weeks or 5 half-lives (whichever is longer).
10. HIstory of hypersensitivity to the study drug or to drugs of similar chemical classes.
11. Current use of medication known to be a strong inhibitor, or moderate or strong inducer, of isoenzyme cytochrome P450 CYP3A.
12. Current use of medications that, to a larger extent, are BCRP, OATP1B1, and/or OATP1B3 substrates.
13. History of HIV or positive test result at screening.
14. Any surgical or medical condition which may jeopardize the subject in case of participation in the study.

    * Chronic need for supplemental oxygen or invasive or non-invasive respiratory support.
    * Liver failure or clinically significant liver disease or dysfunction as indicated by alanine transaminase (ALT) or aspartate transaminase (AST) greater than 2.5 times the upper limit of normal, bilirubin greater than 1.5 times the upper limit of normal, international normalized ratio (INR) greater than 1.5 in the absence of anticoagulation, or presence of diuretic refractory ascites.
    * Elevation of ALT or AST up to 6 times the upper limit of normal is allowed if elevation is determined to be a consequence of immune dysregulation by the site Principal Investigator and if the elevation has been stable for 3 months prior to enrollment.
    * History of significant renal injury/renal disease severely affecting renal function or presence of impaired renal function as indicated by estimated glomerular filtration rate of less than 30 mL/min/1.73 m2.
15. A positive hepatitis B surface antigen (HBsAg), positive hepatitis B PCR, positive hepatitis C PCR, or positive hepatitis C antibody result at screening.
16. Administration of live vaccines starting from 6 weeks before first dose of study medication
17. Subject has a history of malignancy (except lymphoma) within 3 years before the first dose of study medication or has evidence of residual disease from a previously diagnosed malignancy, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
18. Subject has a previous diagnosis of lymphoma that has been treated with chemotherapy, radiotherapy, or transplant within 1 year of the first dose of study medication or is anticipated to require lymphoma treatment within 6 months of the first dose of study medication.
19. Subject has uncontrolled post-transplant lymphoproliferative disease-like Epstein-Barr virus related lymphoproliferative disease.
20. Donation or loss of 400mL or more of blood within 8 weeks before the first dose of study medication
21. Subject has had major surgery requiring hospitalization or radiotherapy within 4 weeks prior to the first dose of study medication or has a planned or expected major surgical procedure during the study period.
22. Pregnant or nursing (lactating) women.
23. Individuals of child-bearing potential, unless they are using highly effective methods of contraception

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety & Tolerability | From baseline to the end of 24 weeks of treatment
  To assess the number of AEs/SAEs and number of participants with AEs/SAEs

SECONDARY OUTCOMES:
Impact of leniolisib on lymphoproliferation measured as index lesions | From baseline to the end of 24 weeks of treatment
  Percent change from baseline in lymphadenopathy measured as the sum of product of diameters (SPD) in the index lesions selected per the Cheson methodology
Impact of leniolisib on lymphoproliferation measured as non-index lesions | From baseline to the end of 24 weeks of treatment
  Percent change from baseline in lymphadenopathy measured as SPD of measurable non-index lesions selected as per the Cheson methodology
Impact of leniolisib on spleen size | From baseline to the end of 24 weeks of treatment
  Percent change from baseline in splenomegaly measured by three-dimensional (3D) volume and bi-dimensional (2D) size of spleen
Impact of leniolisib on hemoglobin | From baseline to the end of 24 weeks of treatment
  Hemoglobin will be evaluated over time
Impact of leniolisib on platelets | From baseline to the end of 24 weeks of treatment
  Platelet count will be evaluated over time
Impact of leniolisib on neutrophils | From baseline to the end of 24 weeks of treatment
  Absolute neutrophil counts will be evaluated over time
Impact of leniolisib on GLILD or other PID-related ILD | From baseline to the end of 24 weeks of treatment
  The change in CT evidence of GLILD or other PID-related ILD over time will be compared using the Hartmann Scoring Methodology
Impact of leniolisib on pulmonary function in FEV1 | From baseline to the end of 24 weeks of treatment
  Change in FEV1 will be evaluated
Impact of leniolisib on pulmonary function in FVC | From baseline to the end of 24 weeks of treatment
  Change in FVC will be evaluated
Impact of leniolisib on pulmonary function in TLC | From baseline to the end of 24 weeks of treatment
  Change in TLC will be evaluated
Impact of leniolisib on pulmonary function in DLCO | From baseline to the end of 24 weeks of treatment
  Change in DLCO will be evaluated
Impact of leniolisib on B and T cell subsets of interest | From baseline to the end of 24 weeks of treatment
  The percentages of naïve B cells, CD21low B cells, and T regulatory cells over time
Impact of leniolisib on CXCL13 and soluble IL-2Rα levels | From baseline to the end of 24 weeks of treatment
  The levels of CXCL13 and soluble IL-2Rα over time
To assess the PK of leniolisib in CVID (Cmax) | From baseline to the end of 24 weeks of treatment
  PK parameters for leniolisib defined by Cmax
To assess the PK of leniolisib in CVID (AUC0-t) | From baseline to the end of 24 weeks of treatment
  PK parameters for leniolisib defined by AUC0-t
To assess the PK of leniolisib in CVID (Tmax) | From baseline to the end of 24 weeks of treatment
  PK parameters for leniolisib defined by Tmax
To assess the PK of leniolisib in CVID (T½) | From baseline to the end of 24 weeks of treatment
  PK parameters for leniolisib defined by T½

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - National Institute of Health, Bethesda, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Texas Children's Hospital, Houston, Texas
- IIS La Fe, Valencia, Spain
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom